CLINICAL TRIAL: NCT01661179
Title: A Phase I/II, Open-label Study to Evaluate the Safety and Tolerability of Vandetanib 300 mg/Day in Japanese Patients With Unresectable Locally Advanced or Metastatic Medullary Thyroid Carcinoma
Brief Title: Evaluate the Safety and Tolerability of Vandetanib in Japanese Patients With Medullary Thyroid Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00098
Record Dates: First submitted 2012-07-17; First posted 2012-08-09 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Unresectable Locally Advanced or Metastatic, Medullary Thyroid Carcinoma
Keywords: Medullary Thyroid Carcinoma; Medullary Thyroid Cancer; Vandetanib
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Medullary | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vandetanib 300mg (Experimental): 300 mg/day vandetanib
  Interventions: Drug: Vandetanib 300mg

INTERVENTIONS:
Drug: Vandetanib 300mg — 300 mg oral dose once daily (100 mg x 3 tablets)
  Other Names: ZD6474

SUMMARY:
Open-label Study to Evaluate the Safety and Tolerability of Vandetanib 300 mg/day in Japanese Patients with Unresectable Locally Advanced or Metastatic Medullary Thyroid Carcinoma.

DETAILED DESCRIPTION:
A Phase I/II, Open-label Study to Evaluate the Safety and Tolerability of Vandetanib 300 mg/day in Japanese Patients with Unresectable Locally Advanced or Metastatic Medullary Thyroid Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Written consent from female or male Japanese patients aged 20 years and over. Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status.
* Previous diagnosis of unresectable, locally advanced or metastatic, hereditary or sporadic Medullary Thyroid Carcinoma(MTC).
* Patients who have a good overall health status(World Health Organization (WHO) Performance status 0-2).
* Patients who have appropriate renal conditions confirmed by test results for taking part in the study.
* For patients with measurable disease(at least one lesion, not irradiated within 12 weeks of study registration, with longest diameter more or equal 10mm (lymph nodes minimum more or equal 15 mm) with CT or MRI).

Exclusion Criteria:

* Patients with brain metastases or spinal cord compression.
* Patients with significant abnormal ECG (QTcB correction unmeasurable or more than 480 ms)findings and /or significant cardiac conditions or events, uncontrolled hypertension and evidence of severe lung disease.
* Abnormal electrolytes such as potassium, magnesium and calcium, or abnormal organ functions such as decreased creatinine clearance.
* Patients with significant abnormal laboratory findings (to include abnormal liver function tests (bilirubin more than 1.5xULRR, and ALT, AST, or ALP more than 2.5xULRR or 5.0xULRR if related to liver metastases).
* Prior treatment (major surgery, radiation therapy, chemotherapy, or other investigational drugs) received within 28 days before registration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, MD, Study Director — Sanofi
Locations (4):
- Japan (4):
  - Research Site, Fukuoka
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Shinjuku-ku

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=356&filename=D4200C00098_Clinical_Trial_Disclosure_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 12 November 2012 to 18 June 2013, 14 participants were treated by 4 centers in Japan to receive vandetanib.
Pre-assignment Details: 16 participants were screened; 14 participants were treated.
Groups:
- Vandetanib 300 mg: Vandetanib at 300 mg using 3 x 100 mg vandetanib tablets were dosed orally, once daily
Period: Overall Study
Arm/Group | Vandetanib 300 mg
Started | 14
Completed | 8
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other Eligibility criteria | 4

BASELINE CHARACTERISTICS:
Arm/Group | Vandetanib 300 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (10.21) [37 to 71]
Age, Customized [Number; unit: Participants]
  >=20 - <50 years | 6
  >=50 - <65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Within the First 56 Weeks After the First Dose of Vandetanib
Description: ORR is defined as the percentage of patients who have a confirmed CR (Disappearance of all target lesions) or PR (>=30% decrease in the sum of diameters of target lesions) prior to any evidence of progression as defined by RECIST V1.1. This percentage is calculated with only patients who had at least measurable lesion in the efficacy analysis set.
Time Frame: Sept 2012 to May 2014
Population: All patients with post-baseline efficacy assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vandetanib 300 mg
Number analyzed (Participants) | 13
percentage of participants | 38.5 [13.86 to 68.42]

ADVERSE EVENTS:
Arm/Group | Vandetanib 300 mg
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib 300 mg (N=14)
Ascites (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib 300 mg (N=14)
Chalazion (Eye disorders) | 1 (1)
Corneal opacity (Eye disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Fatigue (General disorders) | 3 (5)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (8)
Anisakiasis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (5)
Haemoglobin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eyelid function disorder (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Keratopathy (Eye disorders) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 11 (17)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Mucosal erosion (General disorders) | 1 (1)
Oedema (General disorders) | 4 (4)
Oedema mucosal (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4)
Paronychia (Infections and infestations) | 3 (3)
Rash pustular (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Blood calcium increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (5)
Renal impairment (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.